# Prevalence of Acute Injuries in Amateur and Elite Mountain Bikers

Study Type: Complete anonymous questionnaire Study Design: Cross-sectional observational study

Study Categorisation: N/A

Study Registration: ClincialTrials.gov

NTC03690219

Sponsor: Thim van der Laan, Thim van der Laan AG,

Weststrasse 8, 7302 Landquart

+41 81 300 01 70

Principal Investigator: Dr. Ron Clijsen, PhD

University of Applied Sciences of Southern Switzerland SUPSI,

Rehabilitation and Exercise Science Laboratory (RESlab),

Weststrasse 8, 7302 Landquart

+41 81 300 01 75

Protocol ID According to Article 25 of the Human Research Ordinance, this

anonymous questionnaire does not require ethics approval.

Protocol Version and Date: Version 01 (dated xxx)

### CONFIDENTIAL

The information contained in this document is confidential and the property of the sponsor. The information may not - in full or in part - be transmitted, reproduced, published, or disclosed to others than Regulatory Authority(ies) without prior written authorisation from the sponsor except to the extent necessary to obtain informed consent from those who will participate in the study.

#### 1. Introduction

Mountain biking has developed into a popular sport performed by both amateurs and professionals. Physical activity is often related to an increasing risk of injury which may lead to high socioeconomic costs. To avoid accident-related injuries, each racing discipline demands its own set of specific skills and training regimens. The aim of this study is to perform a descriptive analysis of the causes and effects of mountain biking related injuries in amateur and professional athletes.

#### 2. Methods

A survey (as outlined below) of mountain biking related injuries will be conducted on the participants of the Swiss Epic mountain bike event in 2017 held in Valais. The retrospective questionnaire is designed in accordance with existing literature ((Gaulrapp et al., 2001; Lareau and McGinnis, 2011), will include 25 questions and will be translated into English, French, Italian, Spanish and German. The participants will be asked to tick the most appropriate answer. The questionnaire aimes to assess the athletes' 1) basic demographics, riding level and years of experience, 2) number of races per year and mean hours of training per week, 3) number and kind of suffered injuries related to mountain biking and medical treatment requirement, 4) and amount and kind of protective gear items.

## 3. Statistical analysis plan

Data analyses will be performed using the Statistical Package for Social Sciences (SPSS), version 24.0 (IBM Corporation, Armonk, NY, USA).

Descriptive statistics [means  $\pm$  standard deviations (SD) and relative frequencies (%)] will be retrieved. Pearson correlations will be used to assess correlations between the outcome variables. Chi-squared tests will be applied to determine group differences of injury prevalence and the occurrence of severe, respectively mild injury events. Multivariate logistic regressions will be performed to evaluate predictive factors among the outcome variables (independent variables) of severe injury events (dependent variable; no severe injury = 0 versus severe injury = 1) in elites and amateurs separately. Independent samples t-tests will be used to evaluate mean group differences in demographics, and training and injury related variables between the elite and the amateur mountain bikers. P-values < 0.05 will be considered as statistically significant. According to Cohen (1992), effect sizes will be calculated for the correlation analyses and defined as follows; r = 0.20 small, r = 0.50 medium, r = 0.80 strong.







# **Mountain biking Injury Questionnaire**

Thank you for agreeing to take part in this important questionnaire about mountain biking injuries. The information we can obtain from this survey may help to improve the knowledge about injury prevalence in mountain biking. With this knowledge, it may be possible to improve safety in future and prevent injury.

Be assured that all answers you provide will kept in the strictest confidentiality. This survey is anonymous. Do not write your name on the survey.

Please tick only the most correct answer.





University of Applied Sciences and Arts of Southern Switzerland

| Gender | | | Date of birth | |
|---|---|---|---|---|
| ☐ male | ☐ female | □ other | | (day/month/year) |
| Race format | | | | |
| □ swiss epic □ swiss epic flow | ☐ swiss epic 2 day ☐ swiss epic 2 day flow | | | |
| | years do you participa | nte in mountain biking? | | |
| Years | | | | |
| 2. On what level do | you participate in mou | untain biking? | | |
| ☐ recreational | □ amateur | □ elite-amateur | ☐ professional | |
| 3. What's your moti | vation to participate in | n mountain biking? | | |
| □ risk | □ challenge | ☐ health factor | □ fun | $\square$ beeing outdoors |
| □ excitement | ☐ physical exercise | • | | |
| 4. Rider type | | | | |
| ☐ cross country | ☐ trail riding | ☐ all mountain | ☐ downhill | ☐ freeride |
| 5. Pedal System | | | | |
| □ cleat (i.e. Shimano SPD) | | □ platform | | |
| 6. Estimated training | g hours per week in re | egard to the season | | |
| Spring<br>h/Week | Summer<br>h/Week | Autumn<br>h/Week | <i>Winter</i><br>h/Week | |
| 7. How many races | per year | | | |
| 8. Protective gear | | | | |
| ☐ helmet | ☐ gloves | □ eyewear | ☐ upper armour | ☐ lower armour |
| □ other | | | | |
| 9. Number of injurie | s obtained during mo | untain biking | | |
| 10. How long ago wa | s your most recent inj | ury? | | |
| 11. Mechanism of inj | urv | | | |
| □ loss of control | □ loss of traction | ☐ collision with o | bject □ collision with | n rider |
| □ unknown | □ other | | | |







| 12. Se | verity of injury (i | f more than one injury oc | ccurred, choose the most | severe one) | |
|---|---|---|---|---|---|
| | medical<br>nent needed | ☐ self-administrated medical treatment | ☐ MD administrated medical treatment | ☐ Medical treatment in ER | ☐ Overnight hospitalization |
| 13. Bo | dy location affec | eted | | | |
| □ har | nd/finger | $\square$ calf and knee | $\square$ hip and thigh | ☐ trunk | $\square$ foot and ankle joints |
| □ sho | oulder | □ head | ☐ internal organs | $\square$ upper arm and forearm | |
| 14. Ty | pe of injury | | | | |
| □ bor | ne fractures | ☐ joint injuries | $\square$ skin and soft tissue | sue injuries | |
| 15. Da | ys return to spo | rts | | | |
| | | days | | | |
| 16. Da | ys return to worl | k | | | |
| | | days | | | |
| 17. Dic | d you fully recov | er from the injury? | | | |
| ☐ full | recovery | ☐ partial recovery | | | |
| 18. Do | you experience | injury related pain befo | ore/during/after mounta | in biking? | |
| □ bef | ore | ☐ during | □ after | □ no | |
| 19. Do | you experience | NOT injury related pair | n before/during/after mo | ountain biking? | |
| □ bef | ore | ☐ during | □ after | □ no | |
| 20. If y | ou experience N | IOT injury related pain, | where is it located? | | |
| □ kne | ee | □ neck | ☐ lower back | □ hip | □ buttocks |
| □ oth | er | | | | |
| 21. Tre | eatment of musc | le soreness/problems | | | |
| □ ma | ssage lotions | $\square$ electrostimulation | ☐ supplements | ☐ NSAID pain reliefers | |
| □ coc | oling applications | | □ other | (i.e. Ibuprofen, dafa | algan, aspirin, voltaren) |
| 22. Do | you use warmin | ng up cremes/ointments | s before the race? | | |
| □ yes | 3 | □ no | | | |
| 23. Do | you use any cre | emes/ointments after th | e race? | | |
| □ yes | 3 | □ no | | | |
| 24. Do | you use any Pe | rskindol products? | | | |
| □ yes | 3 | □ no | | | |
| 25. If y | ves, before/durin | g/after race? | | | |
| □ bef | ore | ☐ during | □ after | | |

Mountain biking Injury Questionnaire